CLINICAL TRIAL: NCT02320734
Title: A Randomized Controlled Double-blinded Trial Comparing the Effect of on Demand vs Deep Neuromuscular Relaxation on Rating of Surgical and Anesthesia Conditions in Patients Undergoing Thoraco-laparoscopic Esophagectomy
Brief Title: Deep Neuromuscular Relaxation in Patients for Thoraco-laparoscopic Esophagectomy
Acronym: DEPTH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, D.P.Veelo, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2014-211; 2014-002147-18 (EudraCT Number); MISP51412 (Other Grant/Funding Number: Merck Sharp & Dohme BV)
Record Dates: First submitted 2014-12-12; First posted 2014-12-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Neuromuscular Block; Esophageal Cancer; Surgery
Keywords: surgical rating scale; neuromuscular relaxation; Anaesthesia; minimally invasive esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deep neuromuscular relaxation (Active Comparator): continuous infusion of rocuronium 0.6 mg/kg/hr (group 1). On demand bolus rocuronium can be given if demanded by anesthesiologist or surgeon
  Interventions: Drug: Rocuronium
- on demand neuromuscular relaxation (No Intervention): continuous infusion of NaCl 0.9% 0.06 ml/kg/hr (group 2) On demand bolus of Rocuronium will be given when demanded by anesthesiologist or surgeon.

INTERVENTIONS:
Drug: Rocuronium — Rocuronium given continuously to reach deep neuromuscular block
  Other Names: Esmeron
  Arms: deep neuromuscular relaxation

SUMMARY:
Rationale: Endoscopic (thoraco-laparoscopic) esophageal surgery is a high risk procedure where the use of deep neuromuscular block (NMB) may increase field visibility and anaesthesia conditions. Under these conditions, boluses of muscle relaxants can be given on indication only OR by continuous infusion. We hypothesize that deep NMB by continuous infusion of rocuronium as compared to on demand bolus administration facilitates surgical and anesthesia conditions during thoraco-laparoscopic esophageal resection but higher doses of sugammadex are needed to reverse NMB at the end of surgery.

Objective: Primary objective is to evaluate the use of deep muscle relaxation versus on indication only on surgical and anesthesia conditions in patients for endoscopic esophageal resection. Secondary objectives are to evaluate the (hypothetical) dose of sugammadex needed in both groups in an economical perspective and to compare the intra-operative cardiac and respiratory incidents and post-operative complication rate of both groups.

Study design: a single-center randomized controlled double-blinded intervention study.

Study population: All patients > 18 years to undergo a thoracolaparoscopic esophageal resection.I Intervention: Patients are randomized to receive either continuous infusion of rocuronium 0.6 mg/kg/hr (group 1) or continuous infusion of NaCl 0.9% 0.06 ml/kg/hr (group 2). On demand boluses of Rocuronium 0.3 mg/kg can be given in both groups.

Main study parameters/endpoints: The primary outcome parameter of this study is the SRS during the abdominal phase of thoracolaparoscopic esophageal surgery. Secondary outcomes measured are SRS during the thoracic phase, the number of on demand boluses infused, the dose of Sugammadex needed in both groups to reach a TOF of > 90%, duration of surgery, a cost-analysis, the incidence of intra-operative cardiac and respiratory incidents and the ability of surgeons to estimate which neuromuscular blocking regime was given to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients, undergoing elective thoraco-laparoscopic esophageal resection (either Ivor Lewis or McKeown variant)
* Written informed consent

Exclusion Criteria:

* pregnancy
* Known allergies for aminosteroid-type muscle relaxants or sugammadex.
* Severe kidney dysfunction (GFR < 30), patients on dialysis
* Liver function disorders
* Myasthenia Gravis or other (neuro)muscular diseases
* Patients with carcinomatosis
* Use of anti-epileptics and lithium or drugs containing Kinin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rating of surgical conditions (SRS) during the abdominal phase of the operation. | during operation

SECONDARY OUTCOMES:
Rating of SRS during thoracic phase of the operation. | during operation
Number of on demand boluses infused, indication of on demand bolus administration | during operation
Rating of anesthesia conditions | during operation
  peak and mean respiratory pressure, incidence peak insufflation pressure >35 mmHg. Depth of NBM at the end of surgery. Time until spontaneous breathing, time until extubation. Peroperative cardiac and respiratory incidents, peroperative surgical complications.Tiem to reversal of NMB, % of recurarisation
Costs (euro's) associated with use of Rocuronium, Sugammadex, operation time and length of stay ICU. | during operation and an average of 4 weeks thereafter
  amount of rocuronium used (mg); Dose of sugammadex needed (mg), duration of surgery, hypothetical need for post-operative ventilation if sugammadex would not be available(%).
Number of correct estimates of group randomization by surgeons | directly after operation
  Surgeons will guess in which group the patient was randomized (%) and the reason for this choice will be registrated. Accordingly we can estimate whether the surgeons complaints of inadequate NMB are justified and additionally, the chance of bias affecting main outcome parameter.

OTHER OUTCOMES:
length of stay ICU/PACU | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
need for re-intubation | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
post-operative surgical complications | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
VAS-scores | 24-hours post operation
Abdominal and thoracic insufflation pressures | During operation

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, prof, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Denise P Veelo, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Veelo DP, Gisbertz SS, Binnekade JM, Hannivoort RA, Bosman JA, Geerts BF, Blobner M, van Berge Henegouwen MI, Hollmann MW. On-demand versus continuous rocuronium infusion for deep neuromuscular relaxation in patients undergoing thoraco-laparoscopic esophagectomy: a randomized-controlled clinical trial (DEPTH). Can J Anaesth. 2019 Sep;66(9):1062-1074. doi: 10.1007/s12630-019-01373-0. Epub 2019 Apr 25. PMID 31025258
- [Derived] Veelo DP, Gisbertz SS, Hannivoort RA, van Dieren S, Geerts BF, van Berge Henegouwen MI, Hollmann MW. The effect of on-demand vs deep neuromuscular relaxation on rating of surgical and anaesthesiologic conditions in patients undergoing thoracolaparoscopic esophagectomy (DEPTH trial): study protocol for a randomized controlled trial. Trials. 2015 Aug 5;16:331. doi: 10.1186/s13063-015-0849-0. PMID 26242177